CLINICAL TRIAL: NCT06232694
Title: Clinical Study Protocol of Idarubicin, Cytarabine, and Venetoclax -Induced Remission Followed by Consolidation Therapy With Medium-dose Cytarabine Combined With Venetoclax in Newly Diagnosed Adult Acute Myeloid Leukemia
Brief Title: Clinical Study Protocol of IAV-induced Remission Followed by Consolidation Therapy With MDCyta+Ven in ND-AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Huai'an First People's Hospital (Other); Yancheng First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-508
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Administration, Oral; Idarubicin; Infusions, Intravenous; Cytarabine; Injections, Subcutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction therapy and consolidation therapy after remission (Experimental): Induction therapy:Venetoclax + idarubicin + cytarabine Consolidation therapy after remission:Venetoclax + cytarabineIf The patient meets the criteria for autologous hematopoietic stem cell transplantation (ASCT) during the treatment process, they can undergo ASCT.If the patient meets the criteria for transplantation and there is a suitable donor, they can undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT).
  Interventions: Drug: Venetoclax : 100mg on day 1, 200mg on day 2, 400mg on days 3 to 8; oral administration;; Drug: Venetoclax (Venetoclax): 400mg on day 1 to day 7; oral administration;; Other: utologous stem cell transplantation (ASCT) /allogeneic hematopoietic stem cell transplantation (allo-HSCT).

INTERVENTIONS:
Drug: Venetoclax : 100mg on day 1, 200mg on day 2, 400mg on days 3 to 8; oral administration; — Induction Phase Regimen
  Other Names: Idarubicin (Idarubicin): 10-12mg/m2 on days 1 to 3; intravenous infusion; ;Cytarabine (Cytarabine): 100mg/m2 on days 1 to 7; intravenous infusion or subcutaneous injection.
Drug: Venetoclax (Venetoclax): 400mg on day 1 to day 7; oral administration; — Consolidation therapy after remission
  Other Names: Cytarabine: 2g/m2 every 12 hours on day 1 to day 3; intravenous infusion;
Other: utologous stem cell transplantation (ASCT) /allogeneic hematopoietic stem cell transplantation (allo-HSCT). — Four cycles in total.Patients who meet the criteria for autologous stem cell transplantation (ASCT) during the treatment process can undergo ASCT.Patients who meet the transplantation criteria and have a suitable donor can undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT).

SUMMARY:
This study evaluates the efficacy and safety of the combination of idarubicin and cytarabine induction followed by intermediate-dose cytarabine consolidation with venetoclax in the treatment of newly diagnosed adult acute myeloid leukemia (AML).

This study includes the induction and consolidation phases of AML treatment.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, single-arm clinical study aimed at observing and evaluating the effectiveness and safety of idarubicin and cytarabine induction followed by intermediate-dose cytarabine consolidation therapy in newly diagnosed adult AML. The results of this study will help to understand the efficacy and safety of idarubicin and cytarabine combination therapy followed by intermediate-dose cytarabine consolidation in newly diagnosed adult AML, providing guidance for clinical practice.

Acute myeloid leukemia (AML) is a heterogeneous hematopoietic stem/progenitor cell malignancy. The World Health Organization (WHO) defines AML as a myeloid tumor with primitive cells accounting for 20% or more in peripheral blood or bone marrow. It is also the most common acute leukemia in adults and the tenth leading cause of cancer-related deaths worldwide.Treatment for AML consists of induction therapy and consolidation therapy (including chemotherapy and hematopoietic stem cell transplantation (HSCT)).

The most commonly used is the 3+7 regimen. In 2018, our center conducted a retrospective analysis of 242 newly diagnosed AML patients treated with the standard IA regimen, evaluating its efficacy and adverse reactions, and conducting prognostic factor analysis. The study results showed that the CR rate of one course of IA regimen induction therapy was 81.28%; after repeated induction therapy, the CR rate reached 92.34%, confirming that the IA regimen induction therapy has a high CR rate, consistent with many literature reports.

The FDA has approved the combination therapy of Venetoclax and Decitabine/Azacitidine for elderly (>60 years old) newly diagnosed AML patients who are not eligible for intensive chemotherapy. Venetoclax, the first highly selective BCL-2 inhibitor available globally, is a BH3 mimetic that selectively binds to the BCL-2 protein, displacing and releasing pro-apoptotic proteins that were originally bound to BCL-2, effectively inducing apoptosis in tumor cells.

Currently, preclinical studies have confirmed that the combination of idarubicin and cytarabine with venetoclax has a synergistic effect in the anti-tumor treatment of AML. Based on this, the CAVEAT study included 51 newly diagnosed primary or secondary AML patients aged ≥65 years who had not previously received intensive therapy (including AML patients with monosomal karyotype aged ≥60 years). The median age of the patients was 72 years. The treatment regimen for induction and consolidation therapy included idarubicin, cytarabine, and venetoclax (with reduced intensity for idarubicin and cytarabine). The overall response rate (ORR) was 72%, and the median overall survival (OS) was 11.2 months. Compared to secondary AML, patients with primary AML had a longer median OS (31.3 months vs 6.1 months). The most common non-hematologic adverse reactions included febrile neutropenia (55%), sepsis (35%), and diarrhea (35%). These studies suggest that the combination of idarubicin, cytarabine, and venetoclax is safe and tolerable in elderly fit AML patients, and can provide higher remission rates and longer survival. The results of this study also partly confirm the safety of venetoclax in combination with cytarabine and idarubicin for induction chemotherapy in elderly AML patients.

Given the favorable response rates and survival benefits achieved with the combination of VEN and IA in elderly patients with primary AML, we plan to design a prospective, single-arm, multicenter exploratory clinical trial to determine the efficacy and safety of the IA-based induction regimen combined with VEN (IAV regimen) followed by consolidation therapy with intermediate-dose cytarabine and venetoclax in newly diagnosed adult AML patients. This trial aims to provide evidence-based support for novel induction and consolidation treatment strategies for this patient population.

In this study, we also plan to evaluate the efficacy and safety of the combination of idarubicin, cytarabine, and venetoclax as induction therapy followed by consolidation therapy with intermediate-dose cytarabine and venetoclax in newly diagnosed adult AML patients. The aim is to provide a safer and more effective treatment option for these patients.

After signing the informed consent form, young newly diagnosed/eligible AML patients for intensive therapy will undergo various examinations as specified during the screening period. All eligible participants who do not meet the exclusion criteria should be followed up at baseline and on days 1, 3, 5, 7, 9, 11, 13, 15, and 21 during the induction treatment phase, and on days 1 and 21 of each cycle during the consolidation treatment phase. Follow-up visits should also be conducted at the time of withdrawal from the study or at the end of the study for assessment and monitoring.

After signing the informed consent form, young newly diagnosed/fit for intensive therapy AML patients will undergo screening and various tests as specified during the screening period. All eligible participants who do not meet the exclusion criteria will be assessed at baseline and at days 1, 3, 5, 7, 9, 11, 13, 15, and 21 during the induction therapy phase, and on the first and twenty-first day of each cycle during the consolidation therapy phase. Follow-up visits will be conducted at the time of withdrawal/study completion.

Specific treatment plan:

Induction therapy:

Venetoclax: 100mg on day 1, 200mg on day 2, 400mg on days 3-8; oral administration.Idarubicin: 10-12mg/m2 on days 1-3; intravenous infusion.Cytarabine: 100mg/m2 on days 1-7; intravenous infusion or subcutaneous injection.

Consolidation therapy after remission:

Venetoclax: 400mg on days 1-7; oral administration.Cytarabine: 2g/m2 every 12 hours on days 1-3; intravenous infusion.Four cycles in total.Patients who meet the criteria for autologous stem cell transplantation (ASCT) during the treatment process can undergo ASCT.Patients who meet the transplantation criteria and have a suitable donor can undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed primary AML patients. Diagnostic criteria refer to the 2022 WHO classification.
* Age between 18 and 60 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (see Appendix 2).
* Cardiac ultrasound LVEF ≥ 45%.
* Creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula or measured using a 24-hour urine sample).
* Liver function: Aspartate aminotransferase (AST) ≤ 2.5 × ULN*; Alanine aminotransferase (ALT) ≤ 2.5 × ULN*; Total bilirubin ≤ 1.5 × ULN* (*unless considered due to leukemia infiltration).
* Signed informed consent form.

Exclusion Criteria:

* Acute promyelocytic leukemia (APL).
* Relapsed/refractory AML patients.
* AML patients with known involvement of the central nervous system (CNS).
* Known HIV-infected participants (due to potential drug-drug interactions between antiretroviral drugs and venetoclax). HIV testing will be conducted during screening according to local guidelines or institutional standards.Participants with positive hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Non-active carriers of viral hepatitis or participants with low viral hepatitis viral titers after receiving non-prohibited antiviral therapy will not be excluded.
* Participants who have received strong or moderate CYP3A inducers/inhibitors therapy within 7 days prior to starting study treatment.
* Participants with New York Heart Association (NYHA) functional classification > Grade 2. Grade 2 is defined as patients having cardiac disease with no symptoms at rest but experiencing fatigue, palpitations, dyspnea, or angina with ordinary physical activity.
* Participants with chronic respiratory disease requiring continuous oxygen therapy.
* Patients unable to take oral medications or with malabsorption syndrome.
* Presence of uncontrolled systemic infection (viral, bacterial, or fungal).
* Participants who have previously received venetoclax treatment and/or are currently participating in any other study involving investigational drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The composite complete remission rate (CR+CRi) | Four months from the start of initial induction therapy.
  Composite complete remission rate: the proportion of patients who achieve complete remission (CR) and complete remission with incomplete hematologic recovery (CRi) at the end of induction therapy (CR+CRi).• CR is defined as meeting all of the following criteria: ① bone marrow blasts <5%, no circulating or Auer rod blasts; ② no extramedullary disease; ③ ANC ≥1.0 × 109 /L; ④ platelet count ≥100 × 109 /L.• CRi is defined as PLT ≤100 × 109 /L and/or ANC ≤1.0 × 109 /L, with other criteria for CR being met.

SECONDARY OUTCOMES:
The incidence of hematological adverse reactions during induction therapy | Four months from the start of initial induction therapy.
  Adverse reactions are assessed according to the grading criteria for acute and subacute toxicity reactions of anticancer drugs (WHO) (CTCAE 5.0)

OTHER OUTCOMES:
The duration of neutropenia | Four months from the start of initial induction therapy.
  The number of days with an absolute neutrophil count (ANC) below 0.5×109/L.
Minimal residual disease (MRD) | Four months from the start of initial induction therapy.
  In this study, minimal residual disease (MRD) was detected using real-time quantitative PCR and multiparameter flow cytometry techniques, instead of relying on traditional morphological methods to detect leukemia cells below a certain threshold.
Duration of response (DoR) in complete remission (CR) or complete remission with incomplete hematological recovery (CRi) | Four months from the start of initial induction therapy.
  Duration of response (DoR) is the time from the initial achievement of complete remission (CR/CRi) to either relapse or the last follow-up.
Overall survival (OS) | Four months from the start of initial induction therapy.
  Overall survival (OS) is calculated from the successful screening to the time of patient death or the end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided